CLINICAL TRIAL: NCT01068431
Title: Prospective, Randomized Controlled Trial Comparing the Effect of CircAid(R) Juxta-Fit(tm) Versus Trico Bandages in the Treatment of Leg Lymphedema
Brief Title: Short Term Effectiveness Study of Juxta-Fit Versus Trico Bandages in the Treatment of Leg Lymphedema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nij Smellinghe Hosptial (Other)
Responsible Party: Principal Investigator, R.J. Damstra, MD PhD deramtologist, Nij Smellinghe Hosptial
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NS2NL
Record Dates: First submitted 2010-02-03; First posted 2010-02-15 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Lymphedema
Keywords: lymphedema; conservative treatment; compression therapy; interface pressure
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- trico bandage (Active Comparator): Leg lymphedema stage 2-3
  Interventions: Other: bandaging with trico as active controller
- juxta fit compression device (Experimental): leg lymphedema stage 2/3
  Interventions: Other: bandaging with trico as active controller

INTERVENTIONS:
Other: bandaging with trico as active controller — In general non-elastic bandaging is the compression treatment in lymphedema
  Other Names: Trico bandages (BSNmedical)

SUMMARY:
Juxta-Fit is used for compression treatment. Juxta-Fit is an inelastic compression device which can be easily adjusted to the circumference of the limb and is usually used during the maintenance phase of lymphedema treatment. The aim of the study is to assess the effectiveness of Juxta-Fit in the initial treatment phase of leg lymphedema compared to the traditional treatment with Trico bandages in relation to interface pressure and to explore if self-management by Juxta fit is efficient after a short demonstration. Data are collected at 0-2-24 hours

DETAILED DESCRIPTION:
Application of marketed compression systems (Juxta-Fit or Trico bandages) used for treatment by trained specialists with assessment of the interface pressure and volume reduction. For the first two hours, bandages and Juxta fit will be applied by experienced medical staff and the use of the juxta-fit device will be explained to the patient. Thereafter the devices will be removed and patients in the Juxta fit group will apply the device themselves in the treatment. In this second phase after 2 hours, patients may adjust the Juxta-Fit according to their needs and comfort when they feel the device is getting too loose as activity of self-management during 24 hours. The patient will document this in a diary.

Detailed measuring data:

Volumetry:

Measurements after 0h, 2h and 24 h by using classic water displacement apparatus.

Pressure:

Measurements after 0h, 2h (pre and post system change) and 24 h at the B1 region:

* Supine and standing to calculate the Static Stiffness Index (SSI);
* Supine with and without dorsal flexion to calculate the Dynamic Stiffness index (DSI).

Circumference measurement as safety parameter At 5 cm above the upper part of the patella the circumference is measured at 0-2-24 hours to monitor eventual fluids shift.

Questionnaire

- The Visual Analog Scale (VAS) is used at 0 (pre-treatment), 2 and 24 hours to register the comfort of the materials used.

ELIGIBILITY:
Inclusion criteria:

* Gender: male or female
* More than 18 years of age
* Patients with distal lymphedema of the leg requiring multilayer lymphedema bandaging of the leg stage 2/3 (pitting component)
* The patient is able to understand the study and is willing to give written informed consent to the study.

Exclusion criteria:

* Allergy to one of the used materials
* Proximal lymphedema (involvement of thigh, genitalia)
* Severe systemic diseases causing peripheral edema
* Acute superficial or deep vein thrombosis
* Arterial occlusive disease (stadium II, III or IV) Ankle Brachial Pulse Index (ABPI) <0,8
* Local infection in the therapy area
* Auto-immunological disorders or vasculitis
* Use of systemic corticosteroids
* Inability to don, doff, and adjust the Juxta-Fit
* If the ankle circumference around the malleoli is greater than 38cm or if the difference between the arch circumference and the circumference around the base of the toes is greater than 7cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of a device initial made for the maintenance treatment phase, which is now used in the initial treatment phase during 24 hour | short term study during 26 hours

SECONDARY OUTCOMES:
Quality of life (Visual Analog Scale) and number of self-management interventions by the patient in the study group | short term study during 26 hours

CONTACTS AND LOCATIONS:
Overall Officials: RJ Damstra, MD PhD, Principal Investigator — Nij Smellinghe Hospital
Locations (1):
- Nij Smellinghe hospital, Drachten, Provincie Friesland, Netherlands